CLINICAL TRIAL: NCT04924777
Title: Effects of Moderate Physical Activity on Glycemic Control in Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/0929 Zainab Qadri
Record Dates: First submitted 2021-06-11; First posted 2021-06-14 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Resistance Training; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brisk walk (Experimental)
  Interventions: Other: Brisk Walk; Other: Strength training; Other: Aerobic Exercises
- Aerobic Training (Experimental)
  Interventions: Other: Brisk Walk; Other: Strength training; Other: Aerobic Exercises
- Strength Training (Experimental)
  Interventions: Other: Brisk Walk; Other: Strength training; Other: Aerobic Exercises

INTERVENTIONS:
Other: Brisk Walk — 1-Brisk walk for 30 minutes 2-5 days a week 3-3months
Other: Strength training — 1-Strength Training Exercises for 30 minutes. 2-5 days a week 3-3 months
Other: Aerobic Exercises — 1-Aerobic exercises for 30 minutes 2-5 Days a week 3-3months

SUMMARY:
The study design is to determine the effectiveness of moderate physical activity on g;lycemic control in type 2 diabetes mellitus.

DETAILED DESCRIPTION:
To the best of authors knowledge so far the studies have been conducted on different modes of moderate physical activity on glycemic control in type 2 diabetes, current study goal is to evaluate which mode of moderate physical activity has more significant result on glycemic control in type 2 diabetes and is sustainable in Pakistani society according to the socioeconomic status and cost effectiveness of the modes of moderate physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Participants falling in this category would be recruited into the study.
* Male/female
* Diabetic type 2 patients
* Age: 30-70 years
* BMI >25
* Overweight
* Fat % in male> 25
* Fat % in female >35
* HbA1c level more than 48mmol/mol or >6.5%
* Fasting Plasma Glucose level >126 mg/dl (7.0 mmol/l)
* Random Plasma glucose level >200 mg/dl (11.1 mmol/l)
* Physically active ( have no mobility problems)

Exclusion Criteria:

* Participant failing to fall in this category would be excluded of the study.
* Type 1 diabetes
* Insulin dependant type 2 diabetes
* Gestational Diabetes
* Hypertension
* Cigarette smoking
* Cardiovascular Disease
* Cerebrovascular disease
* Cardiopulmonary Disorders
* Cognition Problems
* Peripheral Artery Disease
* Dyslipidemia
* Proliferative or preproliferative retinopathy
* Nephropathy
* Neuropathy

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
HbA1c Levels | 3 months
  Reduction in HbA1c levels

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmad Awan, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No